CLINICAL TRIAL: NCT05989620
Title: Long-Term Development of Muscular Dystrophy Outcome Assessments (GRASP-01-005)
Brief Title: Long-Term Development of Muscular Dystrophy Outcome Assessments
Acronym: GRASP-01-005
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Sponsor
Other Study IDs: HM20027839
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: LGMD1B; LGMD1C; LGMD1D; LGMD1E; LGMD1F; LGMD1G; LGMD1H; LGMD2A; LGMD2B; LGMD2C; LGMD2D; LGMD2E; LGMD2F; LGMD2G; LGMD2I; LGMD2J; LGMD2K; LGMD2L; LGMD2M; LGMD2N; LGMD2O; LGMD2P; LGMD2Q; LGMD2S; LGMD2T; LGMD2U; LGMD2W; LGMD2X; LGMD2Y
Keywords: Muscular Dystrophy; Myotonic Dystrophy; Limb Girdle Muscular Dystrophy; LGMD; LOPD; Late Onset Pompe Disease
MeSH Terms: conditions — Limb-girdle muscular dystrophy, type 1B; Muscular Dystrophy, Limb-Girdle, Type 1C; Muscular Dystrophy, Limb-Girdle, Type 1D; Muscular Dystrophy, Limb-Girdle, Type 1E; Muscular Dystrophy, Limb-Girdle, Type 1F; Limb-Girdle Muscular Dystrophy, Type 1G; Limb-girdle muscular dystrophy type 2A; Limb-girdle muscular dystrophy, type 2B; Limb-girdle muscular dystrophy, type 2C; Sarcoglycanopathies; Limb-girdle muscular dystrophy, type 2E; Limb-girdle muscular dystrophy type 2F; Muscular Dystrophy, Limb-Girdle, Type 2G; Muscular Dystrophy, Limb-Girdle, Type 2I; Muscular Dystrophy, Limb-Girdle, Type 2J; Walker-Warburg Syndrome; Muscular Dystrophy, Limb-Girdle, Type 2L; Muscular Dystrophy, Limb-Girdle, Type 2M; Muscular Dystrophies; Myotonic Dystrophy; Muscular Dystrophies, Limb-Girdle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples will be collected for biomarker development and retained for future research. No clinical diagnosis will be given to patients as part of this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- LGMD, DM2, LOPD

SUMMARY:
This is a 24-month, observational study of up to 1000 participants with Limb Girdle Muscular Dystrophy (LGMD), Myotonic Dystrophy Type 2 (DM2), and late onset Pompe disease (LOPD).

DETAILED DESCRIPTION:
Limb Girdle Muscular Dystrophy (LGMD) comprise a group of disorders made up of over 30 mutations which share a common phenotype of progressive weakness of the shoulder and hip girdle muscles. While the individual genetic mutations are rare, as a cohort, LGMDs are one of the four most common muscular dystrophies.

Myotonic Dystrophy Type 2 (DM2) is a more recently discovered, rare type of myotonic dystrophy. DM2 is inherited in an autosomal dominant pattern and is caused by an unstable CCTG expansion. DM2 affects the muscles and other body systems (e.g. heart and eyes).

Pompe disease is a rare, multisystemic, hereditary disease which is caused by pathogenic variations in the GAA gene. Late onset Pompe disease (LOPD) refers to cases in which hypertrophic cardiomyopathy did not manifest or was not diagnosed at or under the age of 1 year. LOPD is characterized by skeletal muscle weakness which causes mobility problems and impacts the respiratory system.

The overall goal of this project is to extend prior observational studies conducted within the GRASP LGMD network to define the key phenotypes as measured by standard clinical outcome assessments (COAs) for multiple rare types of muscular dystrophy to hasten therapeutic development.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6-50 years at enrollment
2. Clinically affected (defined as weakness on bedside evaluation in a pattern consistent with proximal weakness)
3. Genetic confirmation of a LGMD, DM2, or LOPD
4. FVC above 30% of predicted

Exclusion Criteria:

1. Any other illness that would interfere with the ability to undergo safe testing or would interfere with interpretation of the results in the opinion of the site investigator
2. Participation in a clinical trial receiving an investigational product

Ages: 6 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study seeks to enroll ambulatory individuals aged 6-50 years at enrollment who are clinically affected by LGMD, DM2, or LOPD.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
To explore the suitability and feasibility of the North Star Assessment for LGMD (NSAD) in the muscular dystrophies | Baseline to 24 months
  The NSAD is a functional scale specifically designed to measure motor performance in individuals with LGMD. It consists of 29 items that are considered clinically relevant items from the adapted North Star Ambulatory Assessment and the Motor Function Measure 20 with a maximum score of 54.

SECONDARY OUTCOMES:
To explore the utility of the 100 meter timed test as a clinical outcome assessment in the muscular dystrophies | Baseline to 24 months
  The participant will be asked to complete 4 laps around 2 cones set 25 meters apart, as quickly and safely as possible, walking or running if able. The total time to complete the 4 laps is recorded in seconds.
To explore the utility of the Performance of the Upper Limb 2.0 (PUL 2.0) assessment as a clinical outcome assessment in the muscular dystrophies | Baseline to 24 months
  The PUL 2.0 is a tool designed for assessing upper limb function in persons with neuromuscular disorders. It was developed as a conceptual framework reflecting the progression of weakness and natural history of functional decline in Duchenne Muscular Dystrophy (DMD). There are 22 scored items; a score of 42 indicates the highest level of independent function and 0 the lowest.
To explore the utility of spirometry as a clinical outcome assessment in the muscular dystrophies | Baseline to 24 months
  Spirometry is a breathing assessment comprised of: seated and supine forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), and slow vital capacity (SVC). This assessment is performed using standardized equipment.
To explore the utility of the LGMD-HI questionnaire as a patient-reported outcome measure in the muscular dystrophies. | Baseline to 24 months
  The LGMD Health Index (LGMD-HI) is a disease-specific, patient-reported measure that assesses overall health-related quality of life in LGMD.
To explore the utility of the PROMIS-57 as a patient-reported outcome measure in the muscular dystrophies. | Baseline to 24 months
  The PROMIS-57 is a set of patient-reported measures developed by the NIH. The social health set of questions evaluates general social health by assessing ability to participate in social roles and activities, companionship, satisfaction with social roles and activities, social isolation, and social support.
  The mental health set evaluates general mental health by assessing anxiety, depression, alcohol use, anger, cognitive function, life satisfaction, meaning and purpose, positive affect, psychosocial illness impact, self-efficacy for managing chronic conditions, smoking, and substance use.
  The physical health set evaluates general physical health by assessing fatigue, pain intensity, pain interference, physical function, sleep disturbance, dyspnea, gastrointestinal symptoms, itch, pain behavior, pain quality, sexual function, and sleep related impairment.
To explore the utility of the Domain Delta as a patient-reported outcome measure in the muscular dystrophies | Baseline to 24 months
  The Domain Delta questionnaire is a patient-reported outcome measure that assesses overall health over the previous 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Johnson, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Aggregated and deidentified data will be shared with qualified investigators upon majority approval of the LGMD investigators.

REFERENCES:
- [Background] van de Velde NM, Hooijmans MT, Sardjoe Mishre ASD, Keene KR, Koeks Z, Veeger TTJ, Alleman I, van Zwet EW, Beenakker JM, Verschuuren JJGM, Kan HE, Niks EH. Selection Approach to Identify the Optimal Biomarker Using Quantitative Muscle MRI and Functional Assessments in Becker Muscular Dystrophy. Neurology. 2021 Aug 3;97(5):e513-e522. doi: 10.1212/WNL.0000000000012233. Epub 2021 Jun 23. PMID 34162720
- [Background] Mendell JR, Al-Zaidy S, Shell R, Arnold WD, Rodino-Klapac LR, Prior TW, Lowes L, Alfano L, Berry K, Church K, Kissel JT, Nagendran S, L'Italien J, Sproule DM, Wells C, Cardenas JA, Heitzer MD, Kaspar A, Corcoran S, Braun L, Likhite S, Miranda C, Meyer K, Foust KD, Burghes AHM, Kaspar BK. Single-Dose Gene-Replacement Therapy for Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1713-1722. doi: 10.1056/NEJMoa1706198. PMID 29091557
- [Background] Pozsgai ER, Griffin DA, Heller KN, Mendell JR, Rodino-Klapac LR. Systemic AAV-Mediated beta-Sarcoglycan Delivery Targeting Cardiac and Skeletal Muscle Ameliorates Histological and Functional Deficits in LGMD2E Mice. Mol Ther. 2017 Apr 5;25(4):855-869. doi: 10.1016/j.ymthe.2017.02.013. Epub 2017 Mar 9. PMID 28284983
- [Background] Mendell JR, Rodino-Klapac LR, Rosales XQ, Coley BD, Galloway G, Lewis S, Malik V, Shilling C, Byrne BJ, Conlon T, Campbell KJ, Bremer WG, Taylor LE, Flanigan KM, Gastier-Foster JM, Astbury C, Kota J, Sahenk Z, Walker CM, Clark KR. Sustained alpha-sarcoglycan gene expression after gene transfer in limb-girdle muscular dystrophy, type 2D. Ann Neurol. 2010 Nov;68(5):629-38. doi: 10.1002/ana.22251. PMID 21031578
- [Background] Potter RA, Griffin DA, Sondergaard PC, Johnson RW, Pozsgai ER, Heller KN, Peterson EL, Lehtimaki KK, Windish HP, Mittal PJ, Albrecht DE, Mendell JR, Rodino-Klapac LR. Systemic Delivery of Dysferlin Overlap Vectors Provides Long-Term Gene Expression and Functional Improvement for Dysferlinopathy. Hum Gene Ther. 2018 Jul;29(7):749-762. doi: 10.1089/hum.2017.062. Epub 2017 Jul 13. PMID 28707952
- [Background] Mayhew AG, Cano SJ, Scott E, Eagle M, Bushby K, Manzur A, Muntoni F; North Star Clinical Network for Neuromuscular Disease. Detecting meaningful change using the North Star Ambulatory Assessment in Duchenne muscular dystrophy. Dev Med Child Neurol. 2013 Nov;55(11):1046-52. doi: 10.1111/dmcn.12220. Epub 2013 Aug 5. PMID 23909763
- [Background] Harris E, Bladen CL, Mayhew A, James M, Bettinson K, Moore U, Smith FE, Rufibach L, Cnaan A, Bharucha-Goebel DX, Blamire AM, Bravver E, Carlier PG, Day JW, Diaz-Manera J, Eagle M, Grieben U, Harms M, Jones KJ, Lochmuller H, Mendell JR, Mori-Yoshimura M, Paradas C, Pegoraro E, Pestronk A, Salort-Campana E, Schreiber-Katz O, Semplicini C, Spuler S, Stojkovic T, Straub V, Takeda S, Rocha CT, Walter MC, Bushby K; Jain COS Consortium. The Clinical Outcome Study for dysferlinopathy: An international multicenter study. Neurol Genet. 2016 Aug 4;2(4):e89. doi: 10.1212/NXG.0000000000000089. eCollection 2016 Aug. PMID 27602406
- [Background] James MK, Alfano LN, Muni-Lofra R, Reash NF, Sodhi J, Iammarino MA, Moat D, Shannon K, McCallum M, Richardson M, Eagle M, Straub V, Marini-Bettolo C, Lowes LP, Mayhew AG. Validation of the North Star Assessment for Limb-Girdle Type Muscular Dystrophies. Phys Ther. 2022 Oct 6;102(10):pzac113. doi: 10.1093/ptj/pzac113. PMID 35932452
- [Background] Hunter M, Heatwole C, Wicklund M, Weihl CC, Mozaffar T, Statland JM, Johnson NE. Limb-girdle muscular dystrophy: A perspective from adult patients on what matters most. Muscle Nerve. 2019 Oct;60(4):419-424. doi: 10.1002/mus.26636. Epub 2019 Jul 24. PMID 31298728
- [Background] Arrigoni F, De Luca A, Velardo D, Magri F, Gandossini S, Russo A, Froeling M, Bertoldo A, Leemans A, Bresolin N, D'angelo G. Multiparametric quantitative MRI assessment of thigh muscles in limb-girdle muscular dystrophy 2A and 2B. Muscle Nerve. 2018 Oct;58(4):550-558. doi: 10.1002/mus.26189. Epub 2018 Aug 22. PMID 30028523
- [Background] Willis TA, Hollingsworth KG, Coombs A, Sveen ML, Andersen S, Stojkovic T, Eagle M, Mayhew A, de Sousa PL, Dewar L, Morrow JM, Sinclair CD, Thornton JS, Bushby K, Lochmuller H, Hanna MG, Hogrel JY, Carlier PG, Vissing J, Straub V. Quantitative magnetic resonance imaging in limb-girdle muscular dystrophy 2I: a multinational cross-sectional study. PLoS One. 2014 Feb 28;9(2):e90377. doi: 10.1371/journal.pone.0090377. eCollection 2014. PMID 24587344
- [Background] Murphy AP, Morrow J, Dahlqvist JR, Stojkovic T, Willis TA, Sinclair CDJ, Wastling S, Yousry T, Hanna MS, James MK, Mayhew A, Eagle M, Lee LE, Hogrel JY, Carlier PG, Thornton JS, Vissing J, Hollingsworth KG, Straub V. Natural history of limb girdle muscular dystrophy R9 over 6 years: searching for trial endpoints. Ann Clin Transl Neurol. 2019 May 16;6(6):1033-1045. doi: 10.1002/acn3.774. eCollection 2019 Jun. PMID 31211167
- [Background] Reyngoudt H, Marty B, Boisserie JM, Le Louer J, Koumako C, Baudin PY, Wong B, Stojkovic T, Behin A, Gidaro T, Allenbach Y, Benveniste O, Servais L, Carlier PG. Global versus individual muscle segmentation to assess quantitative MRI-based fat fraction changes in neuromuscular diseases. Eur Radiol. 2021 Jun;31(6):4264-4276. doi: 10.1007/s00330-020-07487-0. Epub 2020 Nov 21. PMID 33219846
- [Background] Reyngoudt H, Smith FE, Caldas de Almeida Araujo E, Wilson I, Fernandez-Torron R, James MK, Moore UR, Diaz-Manera J, Marty B, Azzabou N, Gordish H, Rufibach L, Hodgson T, Wallace D, Ward L, Boisserie JM, Le Louer J, Hilsden H, Sutherland H, Canal A, Hogrel JY, Jacobs M, Stojkovic T, Bushby K, Mayhew A; Jain Clinical Outcome Study for Dysferlinopathy consortium; Straub V, Carlier PG, Blamire AM. Three-year quantitative magnetic resonance imaging and phosphorus magnetic resonance spectroscopy study in lower limb muscle in dysferlinopathy. J Cachexia Sarcopenia Muscle. 2022 Jun;13(3):1850-1863. doi: 10.1002/jcsm.12987. Epub 2022 Apr 3. PMID 35373496
- [Background] Barnard AM, Willcocks RJ, Finanger EL, Daniels MJ, Triplett WT, Rooney WD, Lott DJ, Forbes SC, Wang DJ, Senesac CR, Harrington AT, Finkel RS, Russman BS, Byrne BJ, Tennekoon GI, Walter GA, Sweeney HL, Vandenborne K. Skeletal muscle magnetic resonance biomarkers correlate with function and sentinel events in Duchenne muscular dystrophy. PLoS One. 2018 Mar 19;13(3):e0194283. doi: 10.1371/journal.pone.0194283. eCollection 2018. PMID 29554116
- [Background] Willcocks RJ, Arpan IA, Forbes SC, Lott DJ, Senesac CR, Senesac E, Deol J, Triplett WT, Baligand C, Daniels MJ, Sweeney HL, Walter GA, Vandenborne K. Longitudinal measurements of MRI-T2 in boys with Duchenne muscular dystrophy: effects of age and disease progression. Neuromuscul Disord. 2014 May;24(5):393-401. doi: 10.1016/j.nmd.2013.12.012. Epub 2014 Jan 11. PMID 24491484
- [Background] Burakiewicz J, Sinclair CDJ, Fischer D, Walter GA, Kan HE, Hollingsworth KG. Quantifying fat replacement of muscle by quantitative MRI in muscular dystrophy. J Neurol. 2017 Oct;264(10):2053-2067. doi: 10.1007/s00415-017-8547-3. Epub 2017 Jul 1. PMID 28669118
- [Background] Willcocks RJ, Rooney WD, Triplett WT, Forbes SC, Lott DJ, Senesac CR, Daniels MJ, Wang DJ, Harrington AT, Tennekoon GI, Russman BS, Finanger EL, Byrne BJ, Finkel RS, Walter GA, Sweeney HL, Vandenborne K. Multicenter prospective longitudinal study of magnetic resonance biomarkers in a large duchenne muscular dystrophy cohort. Ann Neurol. 2016 Apr;79(4):535-47. doi: 10.1002/ana.24599. Epub 2016 Feb 19. PMID 26891991
- [Background] Comi GP, Niks EH, Cinnante CM, Kan HE, Vandenborne K, Willcocks RJ, Velardo D, Ripolone M, van Benthem JJ, van de Velde NM, Nava S, Ambrosoli L, Cazzaniga S, Bettica PU. Characterization of patients with Becker muscular dystrophy by histology, magnetic resonance imaging, function, and strength assessments. Muscle Nerve. 2022 Mar;65(3):326-333. doi: 10.1002/mus.27475. Epub 2021 Dec 30. PMID 34918368
- [Background] Batra A, Lott DJ, Willcocks R, Forbes SC, Triplett W, Dastgir J, Yun P, Reghan Foley A, Bonnemann CG, Vandenborne K, Walter GA. Lower Extremity Muscle Involvement in the Intermediate and Bethlem Myopathy Forms of COL6-Related Dystrophy and Duchenne Muscular Dystrophy: A Cross-Sectional Study. J Neuromuscul Dis. 2020;7(4):407-417. doi: 10.3233/JND-190457. PMID 32538860
- [Background] Pane M, Coratti G, Brogna C, Mazzone ES, Mayhew A, Fanelli L, Messina S, D'Amico A, Catteruccia M, Scutifero M, Frosini S, Lanzillotta V, Colia G, Cavallaro F, Rolle E, De Sanctis R, Forcina N, Petillo R, Barp A, Gardani A, Pini A, Monaco G, D'Angelo MG, Zanin R, Vita GL, Bruno C, Mongini T, Ricci F, Pegoraro E, Bello L, Berardinelli A, Battini R, Sansone V, Albamonte E, Baranello G, Bertini E, Politano L, Sormani MP, Mercuri E. Upper limb function in Duchenne muscular dystrophy: 24 month longitudinal data. PLoS One. 2018 Jun 20;13(6):e0199223. doi: 10.1371/journal.pone.0199223. eCollection 2018. PMID 29924848